CLINICAL TRIAL: NCT05164302
Title: Survey on Skin Surface's Temperature Change When Auricular Acupuncture at Jaw Point (LO1) and Tooth Point (LO3) on Heatlhy Volunteer: a Pilot Study
Brief Title: Skin Surface's Temperature Change When Auricular Acupuncture at Jaw Point and Tooth Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Medical Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-VN01002
Record Dates: First submitted 2021-11-26; First posted 2021-12-20 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Auricular Acupuncture
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: 2-arm crossover design, a pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: LO1 point (Tooth) (Experimental): Participant received auricular acupuncture and sham acupuncture at LO1 point in each side of the ear. In each session, temperature of skin surface at the pinna and lower jaw will be recorded.
  Interventions: Procedure: Auricular acupuncture
- Group B: LO3 point (Jaw) (Experimental): Participant received auricular acupuncture and sham acupuncture at LO3 point in each side of the ear. In each session, temperature of skin surface at the pinna and lower jaw will be recorded.
  Interventions: Procedure: Auricular acupuncture

INTERVENTIONS:
Procedure: Auricular acupuncture — Auricular acupuncture is a method for diagnosing and treating physical and psychosomatic dysfunctions by stimulating a specific point in the ear. To conducting this intervention, we use press tack needles to perform auricular acupuncture.

SUMMARY:
Auricular acupuncture is a method for diagnosing and treating physical and psychosomatic dysfunctions by stimulating a specific point in the ear. Some studies prove that the acupoints on the pinna have a corresponding relationship to the areas of the body. Some research also show that acupuncture acupoints on the body can change the temperature of the corresponding area. In our study, we survey the skin surface's temperature change when using auricular acupuncture at jaw point and tooth point in each side of the ear in heatlhy people.

DETAILED DESCRIPTION:
Participants and Methods: A crossover study is conducted by comparing the in skin surface's temperature change before and after applying auricular acupuncture at Jaw point (LO1) and Tooth point (LO3) in each side of the ear in heatlhy volunteer. A total of 70 participants were randomly assigned to 2 group (A and B) and the allocation was 1:1. In group A: participants received auricular acupuncture at tooth point (LO1) three times: Left ear, Right ear and Sham accupunture. Similarly, LO1 point was replaced by LO3 point (Jaw point) for participants in group B. The primary outcome was change temperature of skin surface at the pinna and lower jaw when using auricular acupuncture at points: LO1 and LO3 in each side of the ear. This trial will be performed as 2-arm crossover design, randomized, controlled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer with normal vital signs
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials
* DASS 21 score within normal limits
* BMI: 18.5 - 23 kg/m2

Exclusion Criteria:

* Inappropriate condition for auricular acupuncture due to skin disease (the skin of the acupuncture point is swollen, hot and red)
* Pregnant woman or breastfeeding woman or woman in period
* Other diseases that could affect or interfere with outcomes, including cardiovascular disease, thyroid disorder, facial disease.
* Taking vasodilators or sunscreen in the examined skin areas
* Taking stimulant (alcohol, beer, coffee, tobacco) within 24h
* Massage or cupping therapy or acupuncture in facial area within 24h
* Playing sport within 2h

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change temperature of skin surface at the pinna and lower jaw when using auricular acupuncture at tooth point in each side of the ear | During procedure

SECONDARY OUTCOMES:
Change temperature of skin surface at the pinna and lower jaw when using auricular acupuncture at jaw point in each side of the ear | During procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Hou PW, Hsu HC, Lin YW, Tang NY, Cheng CY, Hsieh CL. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. doi: 10.1155/2015/495684. Epub 2015 Dec 28. PMID 26823672
- [Background] Tsuruoka N, Katayama S, Seki T, Matsunaga T, Iijima R, Haga Y. Focused Ultrasound PC-6 Stimulation Effects on Blood Flow Volume, Skin Temperature, and Coldness of the Finger and Toe. Complement Med Res. 2019;26(6):404-409. doi: 10.1159/000501149. Epub 2019 Jul 5. PMID 31280256
- [Background] Wang D, Ji B, Yan M, Bai H, Sun X, Dai J, Lu Y, Liu Y, You M, Wu J, Ge Y, Su H, Cheng K, Zhao G. Effect of electroacpuncture of Neiguan (PC 6) and Tianquan (PC 2) on skin temperature, blood perfusion, and adrenoceptor response in rats with acute myocardial ischemia. J Tradit Chin Med. 2017 Dec;37(6):794-803. PMID 32188189
- [Background] Guan L, Li G, Yang Y, Deng X, Cai P. Infrared thermography and meridian-effect evidence and explanation in Bell's palsy patients treated by moxibustion at the Hegu (LI4) acupoint: Overall regulation or a specific target? Neural Regen Res. 2012 Mar 25;7(9):680-5. doi: 10.3969/j.issn.1673-5374.2012.09.007. PMID 25745463